CLINICAL TRIAL: NCT00414505
Title: Korea Institute of Oriental Medicine
Brief Title: A Randomized Controlled Double Blinding Study of Intradermal Acupuncture Treatment on Obesity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wonkwang University (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K06070
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Device: Intradermal Acupuncture Treatment

SUMMARY:
The purpose of this study is to determine whether intradermal acupuncture is effective and safe in the treatment of obesity.

DETAILED DESCRIPTION:
Recently the Studies of auricular acupuncture or Common Acupuncture on obesity have been conducted. Saam acupuncture, the Korean unique acupuncture, is famous with its high efficacy but not established by the scientific way yet. Thus, we tried a double-blind study on the effect of sa-am acupuncture on obesity using intradermal acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* BMI>25, regular menstruation, volunteer

Exclusion Criteria:

* symptomatic obesity, acupuncture treatment within 3 months, >120kg, pregnancy or breast-feeding, hemophilia, dementia, mental illness, arrhythmia, liver cirrhosis, renal failure, pace maker, diabete mellitus, tuberculosis, steroid taker,

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-08; Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Bio-body impedance methods

SECONDARY OUTCOMES:
Cholesterol, Triglycerides, HDL LDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Sung-chul Kim, Ph.D., Study Director — Dept. of Acupuncture & Moxibustion, Wonkwang University Hospital
Locations (1):
- Wonkwang University Hospital, Gwangju, South Korea